CLINICAL TRIAL: NCT06139328
Title: Randomised Study for Double-blind, Placebo-controlled Evaluation of a Single Intravenous Infusion of BI 765845 and Partially-blinded Evaluation of a Single Bolus Administration of BI 765845 on Top of Standard of Care in Patients With Acute Myocardial Infarction
Brief Title: IRI-EXPLORE: A Study to Test Whether BI 765845 Helps People Who Have Had a Heart Attack
Acronym: IRI-EXPLORE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1478-0002; U1111-1291-6320 (Other: WHO/UTN); 2022-502788-39-00 (Other: CTIS)
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sponsor team is also masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- BI 765845 very low dose group, administration type 1 (Experimental)
  Interventions: Drug: BI 765845
- BI 765845 low dose group, administration type 1 (Experimental)
  Interventions: Drug: BI 765845
- BI 765845 medium dose group, administration type 1 (Experimental)
  Interventions: Drug: BI 765845
- BI 765845 high dose group, administration type 1 (Experimental)
  Interventions: Drug: BI 765845
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 765845
- BI 765845 low dose group, administration type 2 (Experimental)
  Interventions: Drug: BI 765845
- BI 765845 high dose group, administration type 2 (Experimental)
  Interventions: Drug: BI 765845

INTERVENTIONS:
Drug: BI 765845 — BI 765845
  Arms: BI 765845 high dose group, administration type 1; BI 765845 high dose group, administration type 2; BI 765845 low dose group, administration type 1; BI 765845 low dose group, administration type 2; BI 765845 medium dose group, administration type 1; BI 765845 very low dose group, administration type 1
Drug: Placebo matching BI 765845 — Placebo matching BI 765845
  Arms: Placebo group

SUMMARY:
This study is open to adults aged 18 and over who have just had a heart attack. The purpose of this study is to find out whether a medicine called BI 765845 helps people who have had a heart attack. The investigators also want to test how well different doses of BI 765845 work and how they are tolerated by people who have had a heart attack.

Participants are randomly assigned to receive either BI 765845 or placebo. Placebo treatments look like BI 765845 treatments but do not contain any medicine. Participants are about 3 times as likely to receive BI 765845 than placebo.

Participants are in the study for 3 months. During this time, they visit the study site 7 times and get 3 phone calls from the site staff. At the visits, the doctors use clinical tests to check the health of the heart. The results are compared between the BI 765845 and placebo groups to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years (or legal age as per local regulations) at the time of signing informed consent
2. Signed and dated written informed consent in accordance with ICH Good Clinical Practice (GCP) and local legislation prior to admission to the trial.
3. Male or female participants of non-childbearing potential. Male participants must be ready and able to use highly effective methods of birth control per ICH M3 (R2) for at least 5 days following investigational medicinl product (IMP) administration. Women who are not of childbearing potential are considered those that fulfil at least one or more of the following: aged 50 years or above and being naturally amenorrhoeic for at least 1 year (amenorrhoea following cancer therapy or during breast-feeding does not rule out childbearing potential) OR have premature ovarian failure confirmed by a gynaecologist OR have undergone bilateral salpingo-oophorectomy OR have undergone hysterectomy OR are affected by Turner syndrome OR have uterine agenesis
4. Onset of symptoms of myocardial ischaemia or myocardial infarct, according to patient report, within a duration of:

Part A: ≥1 hour (h) and ≤12 h prior to randomisation Part B: ≥1 h and ≤12 h prior to randomisation Further inclusion criteria apply.

Exclusion Criteria:

1. Women of childbearing potential
2. Patients indicated for rescue PCI (i.e. after receiving fibrinolysis)
3. Patients presenting with cardiogenic shock defined as either systolic blood pressure (SBP) ≤90 mmHg persisting despite fluid challenge or inotropes/vasopressors use to maintain SBP >90 mmHg.
4. Known history of symptomatic heart failure (HF) with left ventricular systolic dysfunction (i.e. HFrEF) based on verbal medical history as reported by a trial participant or authorised representative
5. Known history of myocardial infarction (MI) with the exception of the index event (based on verbal medical history as reported by a trial participant or authorised representative)
6. Previous coronary artery bypass grafting (CABG) (based on verbal medical history as reported by a trial participant or authorised representative) Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Infarct size measured as the percentage of left ventricular mass that is infarcted as detected using late gadolinium enhancement (LGE) by cardiac magnetic resonance (CMR) | At Day 5

SECONDARY OUTCOMES:
Infarct size measured as the percentage of left ventricular mass that is infarcted as detected using Late gadolinium enhancement (LGE) by cardiac magnetic resonance (CMR) | At Day 90
Difference in myocardial Infarct size (IS) | At Day 5 and Day 90

CONTACTS AND LOCATIONS:
Locations (53):
- Australia (2):
  - South Western Sydney Local Health District, Liverpool, New South Wales
  - The Northern Hospital, Epping, Victoria
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Czechia (3):
  - St. Anna Hospital, Brno
  - University Hospital Brno, Brno
  - General University Hospital, Prague
- Germany (10):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen
  - Universität Leipzig, Leipzig
  - Helios Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein GmbH, Ludwigshafen
  - Universitätsklinikum Ulm, Ulm
- Hungary (3):
  - Semmelweis University, Budapest
  - University of Pecs, Pécs
  - Zala County Hospital, Zalaegerszeg, Zalaegerszeg
- Italy (6):
  - Ospedale San Paolo-Bari-18924, Bari
  - Azienda Ospedaliera Cannizzaro, Catania
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Cona (FE)
  - Osp. Pediatrico Apuano Pasquinucci, Massa
  - A.O. San Gerardo di Monza, Monza
  - Ospedale Mauriziano di Torino, Torino
- Auckland City Hospital, Grafton / Auckland, New Zealand
- Poland (6):
  - American-Polish Heart Clinic, Lesser Poland Cardiovascular Centre, Chrzanów
  - University Hospital in Krakow, Krakow
  - Independent Public Health Care in Myszkow, Myszków
  - University Clinical Hospital in Opole, Opole
  - Independent Public Health Care Center of the Ministry of the Interior in Rzeszow, Rzeszów
  - American Heart of Poland Sp. z o.o.-Tychy-44644, Tychy
- Singapore (3):
  - National University Hospital-Singapore-42005, Singapore
  - National Heart Centre Singapore, Singapore
  - Sengkang General Hospital, Singapore
- Slovakia (3):
  - Cardiovascular Diseases institute of Central Slovakia, Banská Bystrica
  - National Institute of Cardiovascular Diseases, Bratislava
  - Cardiocenter Nitra, s.r.o, Nitra
- Hanyang University Medical Center, Seoul, South Korea
- Spain (6):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen De La Macarena, Seville
  - Complejo Hospitalario Universitario de Vigo, Vigo
- Taiwan (2):
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank
  - Leeds General Infirmary, Leeds
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major regulatory authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency